CLINICAL TRIAL: NCT03664726
Title: Delay Discounting as a Target for Self-Regulation in Prediabetes
Brief Title: MINDD 3: Prediabetes and Delay Discounting
Acronym: MINDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leonard Epstein (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor-Investigator, Leonard Epstein, Principal Investigator, State University of New York at Buffalo
Organization: State University of New York at Buffalo (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: UH2DK109543-02 (NIH)
Record Dates: First submitted 2018-04-04; First posted 2018-09-10 (Actual); Results first posted 2022-08-04 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: PreDiabetes
Keywords: Delay Discounting, Episodic Future Thinking
MeSH Terms: conditions — Prediabetic State | interventions — Water Insecurity

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to complete an episodic future or recent thinking task and asked to describe positive events for different time periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Episodic Future Thinking (EFT) & Neutral Narrative (Experimental): Participants will complete an episodic thinking task to generate episodic cues where they will list and describe events for different time periods.The episodic component of the thinking task will occur while the participants are asked to describe what they are imagining about each event (e.g., vacations, weddings, parties, and so forth). EFT participants will list positive future events they are looking forward to and list events that could happen at different general future time points (e.g., 1 month, 2-6 months, 7-12 months). Participants will also be asked to think about a neutral narrative that describes a situation in which changes to their income are neutral or minimal
  Interventions: Behavioral: Episodic Future Thinking; Behavioral: Neutral Narrative
- Episodic Recent Thinking (ERT) & Neutral Narrative (Active Comparator): Participants will complete an episodic recent thinking task to generate episodic cues where they will list and describe events for different time periods. The episodic component of the thinking task will occur while the participants are asked to describe what they are imagining about each event. ERT participants will list positive recent events they enjoyed and list events that happened recently (e.g. 1 - 7 days ago). Participants will also be asked to think about a neutral narrative that describes a situation in which changes to their income are neutral or minimal (e.g. department job transfer).
  Interventions: Behavioral: Episodic Recent Thinking; Behavioral: Neutral Narrative
- Episodic Future Thinking (EFT) & Scarcity Narrative (Experimental): Participants will complete an episodic thinking task to generate episodic cues where they will list and describe events for different time periods.The episodic component of the thinking task will occur while the participants are asked to describe what they are imagining about each event (e.g., vacations, weddings, parties, and so forth). EFT participants will list positive future events they are looking forward to and list events that could happen at different general future time points (e.g., 1 month, 2-6 months, 7-12 months). Participants will also be asked to think about a narrative to induce a scarcity mindset by describing a situation in which changes to their income are negative (e.g. loss of job).
  Interventions: Behavioral: Episodic Future Thinking; Behavioral: Scarcity Narrative
- Episodic Recent Thinking (ERT) & Scarcity Narrative (Experimental): Participants will complete an episodic recent thinking task to generate episodic cues where they will list and describe events for different time periods. The episodic component of the thinking task will occur while the participants are asked to describe what they are imagining about each event. ERT participants will list positive recent events they enjoyed and list events that happened recently (e.g. 1 - 7 days ago). Participants will also be asked to think about a narrative to induce a scarcity mindset by describing a situation in which changes to their income are negative (e.g. loss of job).
  Interventions: Behavioral: Episodic Recent Thinking; Behavioral: Scarcity Narrative

INTERVENTIONS:
Behavioral: Episodic Future Thinking — Participants will be instructed to use their episodic future cues as they engage in different decision making tasks.
  Other Names: EFT
  Arms: Episodic Future Thinking (EFT) & Neutral Narrative; Episodic Future Thinking (EFT) & Scarcity Narrative
Behavioral: Episodic Recent Thinking — Participants will be instructed to use their episodic recent cues as they engage in different decision making tasks.
  Other Names: ERT
  Arms: Episodic Recent Thinking (ERT) & Neutral Narrative; Episodic Recent Thinking (ERT) & Scarcity Narrative
Behavioral: Scarcity Narrative — Participants will read a narrative to induce a scarcity mindset, in which they are asked to imagine a scenario in which they have lost their job and have no current secondary income.
  Other Names: Scarcity
  Arms: Episodic Future Thinking (EFT) & Scarcity Narrative; Episodic Recent Thinking (ERT) & Scarcity Narrative
Behavioral: Neutral Narrative — Participants will read a narrative in which they are asked to imagine a scenario in which they have been transferred between departmental jobs, with little change in salary/commute.
  Other Names: Neutral
  Arms: Episodic Future Thinking (EFT) & Neutral Narrative; Episodic Recent Thinking (ERT) & Neutral Narrative

SUMMARY:
The proposed research will translate research on delay discounting to the prevention of Type 2 diabetes (T2D) in persons with prediabetes. In this study, the investigators will verify target engagement (DD) by examining if EFT improves DD under conditions shown to increase discounting of the future. Prediabetics will be randomized to receive EFT/ERT in a factorial design when experiencing simulated poverty/neutral conditions, respectively. The effects will be measured on DD. The investigators predict that poverty conditions will increase discounting of the future for ERT subjects, but those receiving EFT will show levels of DD similar to levels observed for participants in the wealth condition.

DETAILED DESCRIPTION:
The prevention of Type 2 diabetes in an obese person with prediabetes requires developing a healthier lifestyle. The rational approach for someone with prediabetes would be to eat healthier, be more active, lose weight, and manage their comorbidities. However, preliminary research suggests that individuals with Type 2 diabetes discount the future and engage in behaviors that maximize current pleasure and short-term gain; thus, daily choices needed to improve future health are rare in this population. Delay discounting (DD) describes the choice of smaller immediate versus larger delayed rewards. This behavioral process is related to a wide variety of health choices, ranging from preventive health to behavioral and medical regimen adherence, including regimens used for Type 2 diabetes. The investigators believe that DD provides a target for one type of self-regulation that can improve a wide variety of health behaviors and medical adherence.

Research from our laboratories has shown that episodic future thinking (EFT), a form of prospection which reduces the bias towards immediate gratification, activates brain regions involved in planning and prospection such that future rewards have increased value and the extent of delay discounting is reduced. Cueing individuals to think about future events during inter-temporal decision-making reduces the rate of DD, eating in and outside of the laboratory, and smoking behavior. The overarching goal of this research is to use an experimental medicine approach to translate basic research on DD and EFT into clinical interventions to prevent the transition from prediabetes to a diagnosis of Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Prediabetes: Participants must have a diagnosis of prediabetes within the last 2 years or meet criteria for prediabetes. The American Diabetes Association guidelines defines prediabetes as Fasting Plasma Glucose (FPG) 100-125 mg/dl, 2h glucose 140-199 mg/dl after Oral Glucose Tolerance Test (OGTT), or hemoglobin A1c (HbA1c) approximately 5.7-6.4%.
* Comorbidities: Participants must have a history of comorbid diagnosis such as hypertension and/or hyperlipidemia to participate in the behavioral portion of this study. Hypertension is defined as blood pressure greater than 140/90 on two separate occasions at least one week apart, or medical management for hypertension (i.e. medications including Lisinopril and Diovan). Dyslipidemia is defined by LDL greater than 130 mg/dl, or non-fasting non HDL cholesterol ≥160mg/dL or medical management for dyslipidemia (medications including Niacin, Lovastatin).

Exclusion Criteria:

* Type 2 Diabetes: Individuals will be excluded if they have Type 2 Diabetes.
* Pregnancy: Women who are pregnant or lactating will be excluded from participation.
* Conditions that affect adherence: Participants should not have a condition that would limit participation which include medical conditions that would affect individuals' ability to use the computer for prolonged period of time; leave the individual unable to ambulate; or current diagnoses of an eating disorder (anorexia, bulimia,), unmanaged psychiatric disorder (depression, anxiety, attention deficit hyperactivity disorder (ADHD), schizophrenia), or an intellectual impairment that would impact study adherence.
* Abnormal glucose related to medications: Participants should not be taking medications that would limit participation and cause abnormal glucose levels (e.g. atypical antipsychotic medications or glucocorticoids) including diabetic drugs such as Metformin.
* Unwilling or unable to eat study food: Participants who are unwilling or not able to eat the study food (a PowerBar) will not be able to take part in this study.

Prior participation in similar studies: Individuals who have recently participated in a laboratory study using similar methods may also be excluded.

* Do not meet discounting criteria: Individuals who do not meet discounting criteria (e.g. nonsystematic discounting) on a delay discounting task may be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard H Epstein, Principal Investigator — SUNY University at Buffalo; Warren K Bickel, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (2):
- United States (2):
  - University at Buffalo, Department of Pediatrics, Division of Behavioral Medicine, Buffalo, New York
  - Fralin Biomedical Research Institute, Virginia Tech Carilion, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available

REFERENCES:
- [Derived] Stein JS, Craft WH, Paluch RA, Gatchalian KM, Greenawald MH, Quattrin T, Mastrandrea LD, Epstein LH, Bickel WK. Bleak present, bright future: II. Combined effects of episodic future thinking and scarcity on delay discounting in adults at risk for type 2 diabetes. J Behav Med. 2021 Apr;44(2):222-230. doi: 10.1007/s10865-020-00178-7. Epub 2020 Sep 28. PMID 32989616
- [Derived] Bickel WK, Stein JS, Paluch RA, Mellis AM, Athamneh LN, Quattrin T, Greenawald MH, Bree KA, Gatchalian KM, Mastrandrea LD, Epstein LH. Does Episodic Future Thinking Repair Immediacy Bias at Home and in the Laboratory in Patients With Prediabetes? Psychosom Med. 2020 Sep;82(7):699-707. doi: 10.1097/PSY.0000000000000841. PMID 32868537

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants completed a screening session prior to randomization (n = 149), in which they completed baseline measures of delay discounting and food reinforcement. 78 participants were eligible and randomized
Groups:
- Episodic Future Thinking (EFT) & Scarcity Narrative: Episodic Future Thinking: Participants will be instructed to use their episodic cues as they engage in different decision making tasks
  Narrative: Participants will also be asked to think about a narrative to induce a scarcity mindset by describing a situation in which changes to their income are negative (e.g. loss of job).
- Episodic Future Thinking (EFT) & Neutral Narrative: Episodic Future Thinking: Participants will be instructed to use their episodic cues as they engage in different decision making tasks
  Narrative: Participants will also be asked to think about a neutral narrative that describes a situation in which changes to their income are neutral or minimal (e.g. department job transfer).
- Episodic Recent Thinking (ERT) & Scarcity Narrative: Episodic Recent Thinking: Participants will be instructed to use their episodic cues as they engage in different decision making tasks
  Narrative: Participants will also be asked to think about a narrative to induce a scarcity mindset by describing a situation in which changes to their income are negative (e.g. loss of job).
- Episodic Recent Thinking (ERT) & Neutral Narrative: Episodic Recent Thinking: Participants will be instructed to use their episodic cues as they engage in different decision making tasks
  Narrative: Participants will also be asked to think about a neutral narrative that describes a situation in which changes to their income are neutral or minimal (e.g. department job transfer).
Period: Overall Study
Arm/Group | Episodic Future Thinking (EFT) & Scarcity Narrative | Episodic Future Thinking (EFT) & Neutral Narrative | Episodic Recent Thinking (ERT) & Scarcity Narrative | Episodic Recent Thinking (ERT) & Neutral Narrative
Started | 21 | 20 | 18 | 19
Completed | 21 | 20 | 18 | 19
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Episodic Future Thinking (EFT) & Scarcity Narrative: Episodic Future Thinking: Participants will be instructed to use their episodic cues as they engage in different decision making tasks
  Narrative: Participants will read a narrative to induce a scarcity mindset, in which they are asked to imagine a scenario in which they have lost their job and have no current secondary income.
- Episodic Future Thinking (EFT) & Neutral Narrative: Episodic Future Thinking: Participants will be instructed to use their episodic cues as they engage in different decision making tasks
  Narrative: Participants will read a narrative in which they are asked to imagine a scenario in which they have been transferred between departmental jobs, with little change in salary/commute.
- Episodic Recent Thinking (ERT) & Scarcity Narrative: Episodic Recent Thinking: Participants will be instructed to use their episodic cues as they engage in different decision making tasks
  Narrative: Participants will read a narrative to induce a scarcity mindset, in which they are asked to imagine a scenario in which they have lost their job and have no current secondary income.
- Episodic Recent Thinking (ERT) & Neutral Narrative: Episodic Recent Thinking: Participants will be instructed to use their episodic cues as they engage in different decision making tasks
  Narrative: Participants will read a narrative in which they are asked to imagine a scenario in which they have been transferred between departmental jobs, with little change in salary/commute.
- Total: Total of all reporting groups
Arm/Group | Episodic Future Thinking (EFT) & Scarcity Narrative | Episodic Future Thinking (EFT) & Neutral Narrative | Episodic Recent Thinking (ERT) & Scarcity Narrative | Episodic Recent Thinking (ERT) & Neutral Narrative | Total
Number analyzed (Participants) | 21 | 20 | 18 | 19 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.57 (12.72) | 50.55 (34.45) | 50.61 (10.41) | 52.89 (11.38) | 50.33 (12.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 13 | 16 | 61
  Male | 4 | 5 | 5 | 3 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 19 | 19 | 16 | 19 | 73
  Unknown or Not Reported | 0 | 1 | 2 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 2
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 8 | 6 | 9 | 28
  White | 14 | 11 | 8 | 10 | 43
  More than one race | 1 | 0 | 2 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 18 | 19 | 78
hbA1c [Count of Participants; unit: Participants]
  HbA1c % 5.4-5.6 | 11 | 10 | 10 | 9 | 40
  HbA1c %5.7-6.4 | 10 | 10 | 8 | 10 | 38
Delay discounting [Mean (Standard Deviation); unit: time*indifference point/delay] — Area under the curve (AUC) for delay discounting included time (x-axis) and indifference point (y-axis), or the amount of money at which the immediate and delayed options are approximately equal. Indifference points are a percentage of the max amount (range 0 - 100). AUC adds the calculated areas for each timepoint from the previous timepoint. Ordinal AUC was used as the measure. Ordinal AUC normalizes the horizontal axis time points to have equal distances between them. AUC ranges from 0 (most impulsive, did not choose delay) to 100 (least impulsive, always chose delay).
  time*indifference point/delay
    $100 Delay Discounting | 0.54 (0.16) | 0.49 (0.17) | 0.52 (0.18) | 0.51 (0.20) | 0.51 (0.17)
    $1000 Delay Discounting | 0.61 (0.19) | 0.57 (0.21) | 0.60 (0.23) | 0.59 (0.20) | 0.59 (0.21)
Site Enrollment [Count of Participants; unit: Participants]
  University at Buffalo | 12 | 13 | 11 | 11 | 47
  Virginia Tech Carilon | 9 | 7 | 7 | 8 | 31
Reinforcing Value of Food; Intensity [Mean (Standard Deviation); unit: number of food portions] — Reinforcing value of food, intensity represents the number of pre-specified portions of food a person would consume when the price is $0/per portion. Population: Two participants did not complete the relative reinforcing value of food questionnaire at baseline.
  number of food portions
    number analyzed (Participants) | 20 | 19 | 18 | 19 | 76
    (all) | 9.9 (6.9) | 10.7 (15.1) | 106 (11.7) | 7.4 (7.1) | 9.6 (10.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Delay Discounting
Description: Delay Discounting will be measured using monetary Delay Discounting tasks with $100 as the delayed reward. Delay discounting is assessed using Area Under the Curve (AUC), or time*indifference point/delay. AUC for delay discounting included time (x-axis) and indifference point (y-axis), or the amount of money at which the immediate and delayed options are approximately equal. Indifference points are a percentage of the max amount (range 0 - 100). AUC adds the calculated areas for each timepoint from the previous timepoint. Ordinal AUC was used as the measure. Ordinal AUC normalizes the horizontal axis time points to have equal distances between them. AUC ranges from 0 (most impulsive, did not choose delay) to 100 (least impulsive, always chose delay).
  This is the difference in delay discounting between session 2 and session 1. Larger numbers indicate a decrease in discounting, or less impulsive, while smaller/negative numbers indicate an increase in discounting, or more impulsive.
Time Frame: Delay Discounting will be measured at baseline (session 1) and after receiving EFT/ERT and Scarcity/Narrative (within about 2 weeks)
Measure: Mean (Standard Deviation); unit: time*indifference point/delay
Groups:
- Episodic Future Thinking (EFT) and Neutral Narrative: Episodic Future Thinking: Participants will be instructed to use their episodic cues as they engage in different decision making tasks
  Narrative: Participants will also be asked to think about a neutral narrative that describes a situation in which changes to their income are neutral or minimal (e.g. department job transfer).
- Episodic Recent Thinking (ERT) and Scarcity Narrative: Episodic Recent Thinking: Participants will be instructed to use their episodic cues as they engage in different decision making tasks
  Narrative: Participants will also be asked to think about a narrative to induce a scarcity mindset by describing a situation in which changes to their income are negative (e.g. loss of job).
Arm/Group | Episodic Future Thinking (EFT) & Scarcity Narrative | Episodic Future Thinking (EFT) and Neutral Narrative | Episodic Recent Thinking (ERT) and Scarcity Narrative | Episodic Recent Thinking (ERT) & Neutral Narrative
Number analyzed (Participants) | 21 | 20 | 18 | 19
time*indifference point/delay | -0.002 (0.032) | 0.108 (0.032) | -0.069 (0.034) | 0.035 (0.033)
Statistical Analysis 1: Comparison: Episodic Future Thinking (EFT) & Scarcity Narrative vs Episodic Future Thinking (EFT) and Neutral Narrative vs Episodic Recent Thinking (ERT) and Scarcity Narrative vs Episodic Recent Thinking (ERT) & Neutral Narrative; Test type: Superiority; p = 0.0034, ANOVA — Comparison of differences by group

2. Primary Outcome: Reinforcing Value of Food
Description: Reinforcing value of food was measured using the relative reinforcing efficacy questionnaire in which participants are asked how many portions of food they would purchase at various prices. Intensity is the number of portions they would purchase and consume when the price is $0.
Time Frame: Session 2
Population: Two participants did not complete Reinforcing value measures
Measure: Mean (Standard Deviation); unit: number of food portions purchased at $0
Arm/Group | Episodic Future Thinking (EFT) & Scarcity Narrative | Episodic Future Thinking (EFT) & Neutral Narrative | Episodic Recent Thinking (ERT) & Scarcity Narrative | Episodic Recent Thinking (ERT) & Neutral Narrative
Number analyzed (Participants) | 20 | 19 | 18 | 19
number of food portions purchased at $0 | 9.9 (2.4) | 10.7 (2.5) | 10.6 (2.5) | 7.4 (2.5)
Statistical Analysis 1: Comparison: Episodic Future Thinking (EFT) & Scarcity Narrative vs Episodic Future Thinking (EFT) & Neutral Narrative vs Episodic Recent Thinking (ERT) & Scarcity Narrative vs Episodic Recent Thinking (ERT) & Neutral Narrative; Test type: Superiority; p = 0.76, ANOVA

3. Secondary Outcome: Change in Working Memory Span
Description: Backwards Corsi is a task that assesses visuo-spatial short term working memory. Participants are asked to watch a series of squares on a computer screen and repeat the sequence backwards. This is done several times and the highest number of correctly remembered locations is the span score, with a possible score of 2 - 9 locations total. Span score represents the number of locations that can be recalled backwards. Larger span scores indicate more locations can be remembered and recalled correctly backwards. This is the difference in score between session 2 and session 1. Larger numbers indicate greater change during the experimental manipulation or better working memory, while smaller or negative numbers indicates lower working memory during the experimental manipulation versus baseline. Numbers close to 0 represent little to no change.
Time Frame: Working Memory will be measured at baseline (session 1) and after receiving EFT/ERT Scarcity/Neutral intervention (up to 2 weeks post-baseline)
Population: Five participants did not complete both measures of the spatial span task.
Measure: Mean (Standard Deviation); unit: number of locations
Arm/Group | Episodic Future Thinking (EFT) & Neutral Narrative | Episodic Recent Thinking (ERT) & Neutral Narrative | Episodic Future Thinking (EFT) & Scarcity Narrative | Episodic Recent Thinking (ERT) & Scarcity Narrative
Number analyzed (Participants) | 19 | 17 | 18 | 19
number of locations | 0.05 (0.48) | 0.41 (0.51) | 0.72 (0.49) | 0.16 (0.48)
Statistical Analysis 1: Comparison: Episodic Future Thinking (EFT) & Neutral Narrative vs Episodic Recent Thinking (ERT) & Neutral Narrative vs Episodic Future Thinking (EFT) & Scarcity Narrative vs Episodic Recent Thinking (ERT) & Scarcity Narrative; Test type: Superiority; p = 0.77, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse event data was examined between the initial session and the second session (about 2 weeks).
Arm/Group | Episodic Future Thinking (EFT) & Scarcity Narrative | Episodic Future Thinking (EFT) & Neutral Narrative | Episodic Recent Thinking (ERT) & Scarcity Narrative | Episodic Recent Thinking (ERT) & Neutral Narrative
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20 | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/18 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT03664726/Prot_SAP_000.pdf